CLINICAL TRIAL: NCT04641026
Title: Discovery of Biological Signatures for Cruciferous Vegetable Intake: Integration of the Broccoli- and Host-derived Metabolome and the Microbiome
Brief Title: Discovery of Biological Signatures for Cruciferous Vegetable Intake (Single Serving)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily Ho, Endowed Chair and Director, Linus Pauling Institute Professor, College of Public Health and Human Sciences, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LPI-8343; 2020-67001-31214 (Other Grant/Funding Number: NIFA)
Record Dates: First submitted 2020-10-29; First posted 2020-11-23 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy
Keywords: broccoli sprout; microbiome; cruciferous vegetable

STUDY DESIGN:
Who Masked: Participant
Masking Description: participant is blinded to the presence or absence of deuterium label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Broccoli sprouts (Active Comparator): Subjects will consume one serving (about 1 cup) of broccoli sprouts with breakfast (bagel, cream cheese, and orange juice).
  Interventions: Other: Broccoli sprouts
- Deuterium oxide-labeled broccoli sprouts (Active Comparator): Subjects will consume one serving (about 1 cup) of deuterium oxide-labeled broccoli sprouts with breakfast (bagel, cream cheese, and orange juice).
  Interventions: Other: Deuterium oxide-labelled broccoli sprouts
- Alfalfa sprouts (Placebo Comparator): Subjects will consume one serving (about 1 cup) of alfalfa sprouts with breakfast (bagel, cream cheese, and orange juice).
  Interventions: Other: Alfalfa sprouts
- Deuterium oxide-labeled alfalfa sprouts (Placebo Comparator): Subjects will consume one serving (about 1 cup) of deuterium oxide-labeled alfalfa sprouts with breakfast (bagel, cream cheese, and orange juice).
  Interventions: Other: Deuterium oxide-labelled alfalfa sprouts

INTERVENTIONS:
Other: Broccoli sprouts — Subjects will consume one serving (about 1 cup) of broccoli sprouts with breakfast (bagel, cream cheese, and orange juice).
  Arms: Broccoli sprouts
Other: Deuterium oxide-labelled broccoli sprouts — Subjects will consume one serving (about 1 cup) of deuterium oxide-labelled broccoli sprouts with breakfast (bagel, cream cheese, and orange juice).
  Arms: Deuterium oxide-labeled broccoli sprouts
Other: Alfalfa sprouts — Subjects will consume one serving (about 1 cup) of alfalfa sprouts with breakfast (bagel, cream cheese, and orange juice).
  Arms: Alfalfa sprouts
Other: Deuterium oxide-labelled alfalfa sprouts — Subjects will consume one serving (about 1 cup) of deuterium oxide-labelled alfalfa sprouts with breakfast (bagel, cream cheese, and orange juice).
  Arms: Deuterium oxide-labeled alfalfa sprouts

SUMMARY:
The purpose of this project is to study the molecular and metabolic profiles in human plasma, urine and microbiome composition following the consumption of broccoli sprouts.

DETAILED DESCRIPTION:
The investigators wish to examine metabolic and molecular markers found in blood and in urine after a single dose of sprouts, and evaluate the importance of the gut microbiome on these parameters. Some subjects will receive broccoli sprouts that are grown in deuterium oxide, a commonly used non-toxic, non-radioactive label for vegetables (Tang, Qin et al. 2005), so researchers can identify metabolites in blood and urine that are directly from consumed sprouts. The investigators plan to feed subjects a standardized breakfast and either broccoli sprouts or alfalfa sprouts (control) and look at the presence of metabolites and activity in the blood and urine 3, 6, 24, 48 and 72 hours following intake as well as changes in microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, 18-60 years of age
* Willing to stop taking herbal and phytochemical (plant-based extract or phytochemical) supplements for 1 week prior to and during the study
* Willing to stop cruciferous vegetable and probiotic supplement, food and beverage intake 1 week prior to and during the study
* Willing to complete a 10-day food diary during the study
* Must be able to give written informed consent

Exclusion Criteria:

* Body Mass Index (BMI) <18.5 or >30.0 kg/m2
* Tobacco use, including e-cigarettes, or smoking of any substance (e.g. cannabis) in the past three months
* Pregnancy, breastfeeding, or planning to become pregnant before completing the study
* Engaging in vigorous exercise more than 7 hours per week
* Have a significant acute or chronic illness such as cardiovascular disease, kidney or liver disease, diabetes, thyroid disorder, or radiation or chemotherapy treatment for cancer within the past five years.
* Use of medications to control cholesterol (e.g. statins, cholestyramine) or fat absorption (e.g. orlistat)
* Have had bariatric surgery (e.g. gastric bypass, gastric banding, sleeve gastrectomy, etc.), other gastrointestinal procedure (e.g. cholecystectomy) or disorders (e.g. Crohn's disease, celiac disease, ulcerative colitis)
* Use of oral antibiotic medication within the 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Urine sulforaphane | Baseline, 3, 6, 24, 48 and 72 hours after consuming a single serving of sprouts
  Change in levels of sulforaphane metabolites in urine
Urine sulforaphane metabolites | Baseline, 3, 6, 24, 48 and 72 hours after consuming a single serving of sprouts
  Change in levels of sulforaphane metabolites in urine
Plasma sulforaphane | Baseline, 3, 6, 24, 48 and 72 hours after consuming a single serving of sprouts
  Change in levels of sulforaphane in plasma
Plasma sulforaphane metabolites | Baseline, 3, 6, 24, 48 and 72 hours after consuming a single serving of sprouts
  Change in levels of sulforaphane metabolites in plasma
Stool sample based gut microbiome composition using 16S rRNA gene sequencing | Baseline, 3, 6, 24, 48 and 72 hours after consuming a single serving of sprouts
  Change in stool sample based gut microbiome composition using 16S rRNA gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Emily Ho, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States